CLINICAL TRIAL: NCT06094946
Title: Parturient Satisfaction With Epidural Analgesia During Parturient Controlled Pump
Brief Title: Parturient Satisfaction With Epidural Analgesia by PCEA or Manual Boluses
Status: Not yet recruiting | Type: Observational
Sponsor: Women's Hospital HUS (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Antti Vaananen, Anesthesiologist MD PhD, Helsinki University Central Hospital
Other Study IDs: PCEA_15102023
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Labor Pain
Keywords: epidural analgesia; labour epidural; patient controlled epidural
MeSH Terms: conditions — Labor Pain | interventions — Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Midwife administered boluses: The epidural analgesia is initiated by a manual bolus of the epidural solution (ropivacaine 1 mg/ml fentanyl 2.5 mug/ml) 10 + 10 ml and then continued on-demand by similar boluses until delivery
  Interventions: Drug: Ropivacaine Hydrocloride; Drug: Fentanyl Citrate
- Automated and parturient controlled epidural boluses: The epidural analgesia is initiated by a manual bolus of the epidural solution (ropivacaine 1 mg/ml fentanyl 2.5 mug/ml) 10 + 10 ml and then continued by automated boluses of the same solution (6ml every 40 minutes) with possibility for the parturient to administer 6 ml extra doses with a 20 minute lock-out. Maximum hourly dose 20 ml.
  Interventions: Drug: Ropivacaine Hydrocloride; Drug: Fentanyl Citrate

INTERVENTIONS:
Drug: Ropivacaine Hydrocloride — 1 mg/ml
Drug: Fentanyl Citrate — 2.5 micrograms/ml

SUMMARY:
Those prospective parturients that express that they may want an epidural labour analgesia for their delivery will be informed about the possibility to choose between a pump driven epidural or midwife administered intermittent boluses.

DETAILED DESCRIPTION:
The purpose is to compare parturient and midwife satisfaction with the epidural labour analgesia when epidural analgesia is maintained by an epidural bolus pump (automated mandatory boluses with patient controlled boluses without background infusion) or midwife administered on-demand boluses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Admitted to the delivery hospital with the prospect of vaginal delivery
* On admission when questioned about planned analgesia expresses that may want an epidural analgesia for the planned vaginal delivery
* After reading the study prochure signs the participation (consent) form
* Sufficient command of Finnish or Swedish to facilitate interview

Exclusion Criteria:

* Contraindications for epidural analgesia
* Planned cesarean delivery
* Age under 18 years

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Parturients coming to the delivery hospital (a tertiary delivery hospital with 8000 deliveries per year and 85 % epidural rate) for intended vaginal delivery and requesting epidural analgesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Parturient satisfaction with analgesia | During use of labour analgesia (up to 6 hours)
  Visual analog scale 0-100 mm (0=dissatisfied; 100=maximum satisfaction)

SECONDARY OUTCOMES:
Midwife satisfaction with epidural labour analgesia | During use of labour analgesia (up to 6 hours)
  Visual analog scale 0-100 mm (0=dissatisfied; 100=maximum satisfaction)
Support person's satisfaction with epidural labour analgesia | During use of labour analgesia (up to 6 hours)
  Visual analog scale 0-100 mm (0=dissatisfied; 100=maximum satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Riina Jernman, MD PhD, Study Director — Helsinki University Hospital Women's hospital
Locations (1):
- HUS/Women's hospital dept of anaesthesia, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous data upon reasonable request with accepted study plan from an academic institution can be shared based on case-by-case assessment by the researchers